CLINICAL TRIAL: NCT05884060
Title: Retrospective Electronic Chart Review to Assess the Prevalence of PNH-clones Among Patients Identified With PNH Risk Factors
Brief Title: Retrospective Chart Review Screening Algorithm to Assess the Prevalence of PNH-clones
Status: Completed | Type: Observational
Sponsor: AZ Delta (Other)
Collaborators: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: B1172022000017
Record Dates: First submitted 2023-05-10; First posted 2023-06-01 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: PNH; Thrombosis
Keywords: PNH; Thrombosis; anemia; aplastic anemia; myelodysplastic syndrome (MDS)
MeSH Terms: conditions — Thrombosis; Anemia; Anemia, Aplastic; Myelodysplastic Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- group 1: patients with evidence of haemolysis without obvious cause
  Interventions: Other: No intervention
- group 2: patients with evidence of bone marrow dysfunction (AA, MDS, unexplained cytopenia)
  Interventions: Other: No intervention
- group 3: patients with thrombosis
  Interventions: Other: No intervention
- group 4: patient group that needs to be eliminated from final high risk cohort: patients with cirrhosis, patients wit septic embolisms & embolisation
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No interventions

SUMMARY:
The present study is a non-interventional retrospective chart review study assessing the prevalence of PNH-clones in patients with PNH risk-factors aged ≥14 years and treated at our hospital. The objective of this study is to develop a PNH screening tool on the hospital Electronic Health Record (EHR) system. An algorithm defining PNH risk groups is developed.

DETAILED DESCRIPTION:
Paroxysmal Nocturnal Hemoglobinuria (PNH) is a life-threatening hematological disorder, but with an effective therapy. Prevalence is estimated between 1-5 per million people, often manifested by cardiovascular, gastrointestinal, neurological or haematological symptoms. Referral is therefore typically to several specialists, resulting in PNH underdiagnosis.

This chart review study consists primarily of developing an algorithm to identify a high-risk cohort of potential PNH patients who need treatment from all registered patients, with maximum ability to find relevant cases. Secondly, this cohort will be manually reviewed by clinicians for final screening. The challenge hence is maximizing the ability to find all relevant PNH patients yet limiting the number to ensure manual review is possible.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥14 years of age
* At least 1 record encoded in the General Hospital Delta (AZ Delta) patient database (HiX) between 20 April 2018 and 1 March 2022
* A history or presence of at least one PNH risk factors identified following retrospective screening of electronic patient records

Exclusion Criteria:

* None

Min Age: 14 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Eligible patients will be identified by retrospective screening of the hospital's electronic patients records using data search queries based on ICD-10 codes, lab results, keyword search in questionnaires, medical reports, notes, radiology reports & medical diagnoses corresponding to one of the PNH Risk factors described:
  1. Patients with evidence of haemolysis without obvious cause
  2. Patients with evidence of bone marrow dysfunction
  3. Patients with thrombosis
Sampling Method: Non-Probability Sample
Enrollment: 568 (Actual)
Dates: Start 2018-04-20 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
PNH risk factors translation into query codes that can be interpreted by a computer system for analysis | 2022
  Three main PNH risk sub-cohorts were constructed, representing patients exhibiting PNH risk factors such as hemolytic anemia (group 1), bone marrow dysfunction (group 2) and thrombosis (group 3). To build these sub-cohorts, queries were created using a combination of structured and unstructured electronic health record (EHR) data, including lab results, diagnoses, medication, questionnaire data, text from medical and radiology reports, notes, and Internation Classification Codes (ICD-10). These sub-cohorts were validated by two hematologists who reviewed randomly selected patients, resulting in several iterations and query optimizations.
Number of patients identified with high risk for PNH clone and per type of screening criteria by developing a computational screening algorithm | 2022
  A computational algorithm was employed for a retrospective EHR analysis, to identify high-risk cohorts of potential PNH patients who need treatment from all registered patients, with maximum ability to find relevant cases. Three main PNH risk sub-cohorts were constructed, representing patients exhibiting PNH risk factors such as hemolytic anemia (group 1), bone marrow dysfunction (group 2) and thrombosis (group 3). These sub-cohorts were validated by two hematologists who reviewed randomly selected patients, resulting in several iterations and query optimizations. Sub-cohorts were subsequently merged and refined into high risk cohorts that undergo further analysis and manual review. Two hematologists independently reviewed and rated medical records to achieve a manual risk stratification of the high risk cohorts.

SECONDARY OUTCOMES:
The number of patients at high risk for PNH, categorized by risk factor, across each medical department | 2023
  To increase awareness of PNH risk factors by medical departments that need to consider PNH lab testing

CONTACTS AND LOCATIONS:
Overall Officials: Dries Deeren, MD, Principal Investigator — AZ Delta
Locations (1):
- AZ Delta, Roeselare, West-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: No